CLINICAL TRIAL: NCT02497755
Title: Connection to Care: Pilot Study of a Mobile Health Tool for Patients With Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Amy Bauer, Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47871
Record Dates: First submitted 2015-02-14; First posted 2015-07-14 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile app (Experimental): Participants will install an app on their smartphone to add to their treatment for depression and/or anxiety.
  Interventions: Behavioral: App for smartphone; Device: smartphone

INTERVENTIONS:
Behavioral: App for smartphone — A smartphone app will send psychoeducation and reminders to patients to complete self-report data, will collect passive data, and will provide aggregated information to a provider dashboard.
Device: smartphone

SUMMARY:
This is a pilot feasibility study of a mobile health tool (smartphone app) for primary care patients receiving treatment for depression or anxiety delivered in an integrated primary care-based behavioral health program.

DETAILED DESCRIPTION:
This research is a feasibility pilot study of a smartphone app using mixed methods. The research seeks to answer the question: "Is a mobile health tool for patient self-management feasible, useful, appropriate, and acceptable for patients and care managers for patients with depression or anxiety treated in an integrated primary-care based behavioral health program?"

ELIGIBILITY:
Inclusion Criteria:

* Be part of the Behavioral Health Integration Program for anxiety and/or depression; Must have an iPhone or Android smartphone with a mobile voice calling plan with a US carrier; Fluent in English

Exclusion Criteria:

* Individual unable or unwilling to accept the terms of the Ginger.io terms of Use; Actively suicidal as determined by a healthcare professional; score of 3 on the Patient Health Questionnaire-9 item 9 (which assesses thoughts of self-harm); or documented history of 2 or more prior suicide attempts; Working diagnosis of psychotic disorder, bipolar disorder, dementia, active substance dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Bauer, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington Neighborhood Clinic, Ravenna, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the caseload of a care manager at the UW Ravenna Neighborhood Clinic who were enrolled in the Behavioral Health Integration Program for depression and anxiety. Recruitment letters were mailed between 6/15/2015 and 7/27/2015.
Groups:
- Patient Mobile App Users: Participants installed an app on their smartphone to add to their treatment for depression and/or anxiety. This smartphone app sent psychoeducation and reminders to patients to complete self-report data, collected passive data, and provided aggregated information to a provider dashboard. Participants used the app for at least 4 weeks, with the option to continue use for up to 12 weeks. After 4 weeks, the research coordinator conducted a phone interview on satisfaction with the app.
- Care Manager Dashboard User: The care manager for the patients participating in this study used an online dashboard to monitor patient usage and responses to mobile app assessments (such as the PHQ-9) as part of her clinical workflow. She used this dashboard for the duration of participant involvement in the study (from 6/25/2015 through 9/30/2015).
Period: Overall Study
Arm/Group | Patient Mobile App Users | Care Manager Dashboard User
Started | 18 | 1
Completed | 17 | 1
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patient Mobile App Users: Participants installed an app for smartphone to add to their treatment for depression and/or anxiety. This smartphone app sent psychoeducation and reminders to patients to complete self-report data, collected passive data, and provided aggregated information to a provider dashboard. Participants used the app for at least 4 weeks, with the option to continue use for up to 12 weeks. After 4 weeks, the research coordinator conducted a phone interview on satisfaction with the app.
- Total: Total of all reporting groups
Arm/Group | Patient Mobile App Users | Care Manager Dashboard User | Total
Number analyzed (Participants) | 17 | 1 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | 16 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | 1 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 7 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | 17 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | 0 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | 0 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | 1 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | 16 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | 0 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 1 | 18
Employment Status [Count of Participants; unit: Participants]
  Full time paid employment | 11 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not working by choice | 1 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Student | 3 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unable to work | 2 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
Education [Count of Participants; unit: Participants]
  Bachelor's degree | 10 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Graduate or professional degree | 3 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  High school/GED | 1 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.
  Some college | 3 | NA — Not assessed | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: App Acceptability as Measured by Number of Patient App Users Who Rate App Easy to Use and Time Spent Reasonable
Description: The number of patients who rated the app was easy to use and the amount of time spent using the app as reasonable when asked about app acceptability in a qualitative interview and via a quantitative survey. Specific survey items included "The technology requires little effort to use," "The technology was easy to learn how to use," "The Ginger.io app is easy to use," and "The time required to answer questions in the Ginger.io app is reasonable." All patients who expressed agreement ("Somewhat Agree," "Agree," or "Strongly Agree") to these items and to similar questions in the qualitative interview were included in the count of patients who found the app acceptable.
Time Frame: Four weeks after intervention started
Population: Overall Number of Participants Analyzed (16) is not consistent with numbers provided in the Participant Flow model (17) because one participant did not complete the quantitative survey used in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Mobile App Users
Number analyzed (Participants) | 16
Participants | 16

2. Primary Outcome: App Acceptability as Measured by Number of Care Manager Dashboard Users Who Rate Dashboard Easy to Use and Time Spent Reasonable
Description: The number of care managers who agreed that the app dashboard was easy to use and that the amount of time spent using the app dashboard was reasonable when asked about app acceptability and benefit vs. burden of use with regard to clinical workflow in a qualitative interview.
Time Frame: 8-16 weeks after final patient participant is enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Care Manager Dashboard User
Number analyzed (Participants) | 1
Participants | 1

3. Primary Outcome: App Usefulness as Measured by Number of Patient App Users Who Rate App as Useful
Description: The number of patients who rated the app as useful to them when asked about app usefulness in a qualitative interview and via a quantitative survey. Specific survey items included "This technology is useful." All patients who expressed agreement ("Somewhat Agree," "Agree," or "Strongly Agree") to this items and to similar questions in the qualitative interview were included in the count of patients who found the app acceptable.
Time Frame: Four weeks after intervention started
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Mobile App Users
Number analyzed (Participants) | 16
Participants | 11

4. Primary Outcome: App Usefulness as Measured by Number of Care Manager Dashboard Users Who Rate Dashboard as Useful
Description: The number of care managers who expressed that the app was useful to them with regard to clinical workflow in a qualitative interview.
Time Frame: 8-16 weeks after final patient participant is enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Care Manager Dashboard User
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Technology Acceptability as Measured by the Obtrusiveness Scale for Pervasive Technology (Modified)
Description: The mean total of patient app users' responses to the modified version of the Obtrusiveness Scale for Pervasive Technology, with a mean score of 13-39 indicating that the app is generally perceived as unacceptable/obtrusive, 40-64 indicating neutrality, and 65-91 indicating that the app is generally perceived as acceptable/unobtrusive.
Time Frame: During weeks 3 and 8
Population: Only 3 participants were analyzed at the 8 week point because only 3 participants of the 17 completed the Week 8 survey.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Patient Mobile App Users
Number analyzed (Participants) | 17
units on a scale
  Week 3 | 69.06 [46 to 90]
  Week 8: number analyzed (Participants) | 3
  Week 8 | 80.33 [72 to 90]

6. Secondary Outcome: Patient Satisfaction as Measured by the Ginger.io Product Feedback Survey.
Description: The mean total of patient app users' responses to the Ginger.io product feedback survey, with a mean score of 7-21 indicating satisfaction with the app, 22-34 neutrality, and 35-49 expressing dissatisfaction.
Time Frame: Days 30, 56
Population: Overall Number of Participants Analyzed (13) is not consistent with numbers provided in the Participant Flow model (17) because 4 of the participants did not complete the Day 30 or the Day 56 survey. Only 2 participants were analyzed at the 56 day point because only 2 participants completed the Day 56 survey.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Patient Mobile App Users
Number analyzed (Participants) | 13
units on a scale
  Day 30 | 19.85 [10 to 28]
  Day 56: number analyzed (Participants) | 2
  Day 56 | 13.00 [13 to 13]

7. Secondary Outcome: Patient Use of the App as Measured by Percentage of App Surveys Completed.
Description: The mean percentage of surveys presented to users through the app that were completed by patient app users in their first 8 weeks of using the app. App survey questions included weekly PHQ-9 and GAD-7 scales and daily measures of mood and medication use as well as satisfaction surveys.
Time Frame: Eight weeks after intervention started
Measure: Mean (Full Range); unit: Percentage of surveys completed
Arm/Group | Patient Mobile App Users
Number analyzed (Participants) | 17
Percentage of surveys completed | 60.24 [28 to 98]

8. Secondary Outcome: Care Team Communication as Measured by the Consumer Assessment of Healthcare Providers and Systems (CAHPS) - Communication Scale
Description: The mean total of patient app users' responses to the 6 items in the Consumer Assessment of Healthcare Providers and Systems (CAHPS) - Communication scale, with a mean score of 0-5 indicating that participants never or almost never experienced good communication with their care team, 6-11 indicating that participants sometimes experienced good communication with their care team, 12-17 indicating that patients usually experienced good communication with their care teams, and a score of 24 indicating that patients always experienced good communication with their care team.
Time Frame: Weeks 4 and 8
Population: Only 13 participants were analyzed at the 8 week point because only 13 participants of the 17 completed the Week 8 survey.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Patient Mobile App Users
Number analyzed (Participants) | 17
units on a scale
  Week 4 | 17 [12 to 28]
  Week 8: number analyzed (Participants) | 13
  Week 8 | 16 [12 to 18]

9. Secondary Outcome: Care Process Measures as Measured by the Number and Type of Contacts With Care Manager.
Description: The mean number of Follow-Up contacts between patient and care manager during the 8 weeks following the patient's activation of the app. (Other types of contacts with the care manager include Initial Assessment and Contact Attempt, but neither of these occurred during the time frame of app use.)
Time Frame: Eight weeks after intervention started
Measure: Mean (Full Range); unit: number of contacts
Arm/Group | Patient Mobile App Users
Number analyzed (Participants) | 17
number of contacts | 1.35 [0 to 3]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of participant involvement in the study (from 6/25/2015 through 9/30/2015).
Arm/Group | Patient Mobile App Users | Care Manager Dashboard User
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/1
Other Adverse Events (participants affected / at risk) | 0/18 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No